CLINICAL TRIAL: NCT06703515
Title: Randomized Controlled Trial of Awake Transnasal Laser-assisted Surgery (TNLS) and Microlaryngeal Surgery for Vocal Cord Cyst
Brief Title: Awake Transnasal Laser-assisted Surgery (TNLS) and Microlaryngeal Surgery for Vocal Cord Cyst
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tam Aurora Ka Yue, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTEC-2023-624
Record Dates: First submitted 2024-11-11; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Vocal Cord Cyst
Keywords: Vocal cord cyst; Transnasal laser surgery; Microlaryngeal surgery; Office based laser surgery; Awake laser laryngeal surgery; Trublue laser

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microlaryngeal surgery (MLS) (Active Comparator): For traditional MLS under general anesthesia, after general anesthesia and intubation with microlaryngeal tube, the patient would be positioned on head-ring support for better alignment and access to glottis. A laryngoscope will be inserted transorally under direct vision and suspended. Vocal cord cysts are visualized with microscope, and removed with microsurgery instruments with microflap technique and sent for routine section. After the surgery, the patient is kept nil-by-mouth until fully awake, and is discharged on same day or the next day depending on the post- operative recovery. Patient will be discharged with voice rest for 3 days.
  Interventions: Procedure: Microlaryngeal surgery (MLS)
- Awake transnasal laser-assisted surgery (TNLS) (Experimental): For TNLS, patients are admitted to the day center on the same morning or afternoon of the surgery with fasting prior 6 hours. After local anesthesia application, a 445nm blue laser is introduced via a working channel of bronchoscope and laser ablation of vocal cord cyst is performed. During the operation, patient will receive continuous SpO2 monitoring with regular blood pressure monitoring. After the procedure, patients are kept nil-by-mouth for 2 hours until anesthesia wears off, meanwhile with close observation in day ward with continuous SpO2 monitor for 1 hour. Patients will be discharged on the same day of the procedure, with voice rest for 3 days.
  Interventions: Procedure: Awake transnasal laser-assisted surgery (TNLS)

INTERVENTIONS:
Procedure: Awake transnasal laser-assisted surgery (TNLS) — For TNLS, patients are admitted to the day center on the same morning or afternoon of the surgery with fasting prior 6 hours. After local anesthesia application, a 445nm blue laser is introduced via a working channel of bronchoscope and laser ablation of vocal cord cyst is performed. During the operation, patient will receive continuous SpO2 monitoring with regular blood pressure monitoring. After the procedure, patients are kept nil-by-mouth for 2 hours until anesthesia wears off, meanwhile with close observation in day ward with continuous SpO2 monitor for 1 hour. Patients will be discharged on the same day of the procedure, with voice rest for 3 days.
  Arms: Awake transnasal laser-assisted surgery (TNLS)
Procedure: Microlaryngeal surgery (MLS) — For traditional MLS under general anesthesia, after general anesthesia and intubation with microlaryngeal tube, the patient would be positioned on head-ring support for better alignment and access to glottis. A laryngoscope will be inserted transorally under direct vision and suspended. Vocal cord cysts are visualized with microscope, and removed with microsurgery instruments with microflap technique and sent for routine section. After the surgery, the patient is kept nil-by-mouth until fully awake, and is discharged on same day or the next day depending on the post- operative recovery. Patient will be discharged with voice rest for 3 days.
  Arms: Microlaryngeal surgery (MLS)

SUMMARY:
This is a prospective randomised controlled trial conducted at two tertiary referral hospitals in Hong Kong to compare the clinical and functional outcomes of office-based awake transnasal laser-assisted laryngeal surgery (TNLS) under local anesthesia to traditional microlaryngeal surgery for vocal cord cyst under general anesthesia.

DETAILED DESCRIPTION:
The aim of the study is to prospectively compare the functional and clinical outcomes of TNLS under local anesthesia and MLS under general anesthesia in managing vocal cord cysts.

Office-based awake transnasal laser-assisted surgery (TNLS) has been gaining popularity in treating different laryngeal lesions, with the advantages of avoiding general anesthetic risks and minimizing healthcare-related costs. In addition, the general waiting time for surgeries under general anesthesia in public hospitals is getting longer due to the increasing population and limited resources. The investigators have recently conducted a novel randomized controlled trial in 2021-2022 comparing the functional and cost-effectiveness of traditional microlaryngeal surgery (MLS) under general anesthesia and TNLS for benign laryngeal lesions (vocal cord polyps, nodules, cysts, granuloma and Reinke's edema), and found that TNLS was superior to MLS in terms of length of stay, intraoperative complications, perioperative throat discomfort and hospital costs; while it was equivalent to MLS in terms of functional outcome, operative time and recurrence rate. However, since the previous study's main goal was to compare TNLS to MLS in a macroscopic perspective in terms of functional outcomes and cost-effectiveness, it had included a wide variety of benign laryngeal lesions, and different vocal cord lesions may respond differently to laser surgery.

Vocal cord cyst is a fluid-filled sac inside the vocal cord, with 2 subtypes: 1) Epidermoid cyst due to epithelial inclusion 2) Mucous retention cyst due to glandular ductal obstruction. Vocal cord cysts typically do not resolve with voice therapy, and are traditionally excised with microlaryngeal surgery with microflap technique or marsupialization. In our previous RCT study, subgroup analysis did not show a significant difference of vocal cord cyst recurrence in both TNLS and MLS group. However, the investigators' cohort had a higher overall vocal cord cyst recurrence rate (13.8%) compared to historic cohort rate of 2.2-8.7% , which may be accounted by that the vocal cord cysts were ablated and marsupialized instead of removed in the TNLS group. Nevertheless, a recent case series by Gao and colleagues showed a good functional outcome of awake KTP-laser marsupialization in selected cases. A larger cohort is warranted to compare TNLS to MLS for vocal cord cyst. Therefore, the investigators would like to conduct a randomized controlled trial to compared tradition MLS surgery to TNLS, with hypothesis that TNLS would be non-inferior to traditional microlaryngeal surgery in benign laryngeal lesions, and with its additional benefits on minimization of anesthetic risks and hospital expenses, hopefully to expand its further application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vocal cord cysts
* older than 18-year-old
* able to independently provide consent
* able to tolerate flexible laryngoscopy would be recruited

Exclusion Criteria:

* under 18-year-old
* unable to independently give an informed consent
* unable to tolerate flexible laryngoscopy
* allergic to local anesthesia
* had unfavorable anatomy such as prolapsing epiglottis precluding adequate visualization, extensive lesions and an expected difficult operation as judged by the surgeons
* with pathologies other than vocal cord cyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Voice-Handicap Index (VHI-30) | From enrolment to post-operative 1year
  The primary outcome was to compare the pre- and post-operative Voice-Handicap Index 30 (VHI-30) of TNLS and MLS groups. The VHI-30 is a 30-item self-administered questionnaire, with score range from 0 to 120, and a score of 120 meaning worst voice score. It has been shown to be a reliable measure for voice treatment outcome. It consists of three subscales, namely physical, functional and emotional. It provides an overall measurement of a person's vocal function and how it influences a person's everyday functioning and experience.

SECONDARY OUTCOMES:
Perceptual evaluation of voice | From enrolment to post-operative 1year
  Perceptual evaluation of voice using the GBRAS scale, in which patients would be required to produce sustained vowel and connected speech voice samples. Score range from 0 to 15, with 15 being the worst score. Two experienced speech-language pathologists blinded to the patient's information would rate the audio recordings.
Acoustic voice analysis - Noise-to-Harmonic ratio (NHR) | From enrolment to post-operative 1year
  Acoustic voice analysis will be performed using PRATT program; Noise-to-Harmonic ratio refers to the ratio between periodic and non-periodic components of a speech sound. A lower NHR score may indicate a worse voice outcome.
Acoustic voice analysis - Jitter | From enrolment to post-operative 1year
  Acoustic voice analysis will be performed using PRATT program; Jitter refers to variation of voice frequency.
Acoustic voice analysis - Shimmer | From enrolment to post-operative 1year
  Acoustic voice analysis will be performed using PRATT program; Shimmer refers to variation of intensity of the voice.
Aerodynamic measure of voice | From enrolment to post-operative 1year
  Aerodynamic measure, maximal phonation time (MPT) would be measured by instructing patients to phonate /a:/ sound for as long as possible after maximal inspiration, at a spontaneous, comfortable pitch and loudness level, for three consequent trials.
Visual analog scale (VAS) | From enrolment to post-operative 1year
  In VAS, patients would be asked to self-rate their voice quality on a visual analog scale of 0 (best) to 10 (worst).
Videostroboscopy - Mucosal wave pattern | From enrolment to post-operative 1year
  Videostroboscopy would be conducted on all patients to look for any impaired mucosal wave form.
Videostroboscopy - Vocal fold closure | From enrolment to post-operative 1year
  Videostroboscopy would be conducted on all patients to compare the degree of vocal fold closure.
Procedure-oriented outcomes - Reoperation | From perioperative period to post-operative 1 year
  Comparison of the rate of reoperation for recurrence vocal cord cyst between two groups.
Procedure-oriented outcomes - Disease recurrence | From perioperative period to post-operative 1 year
  Comparison of the rate of vocal cord cyst recurrence between two groups.
Procedure-oriented outcomes - Length of hospital stay | From perioperative period to post-operative 1 year
  Comparison of the length of hospital stay (number of day) between two groups.
Procedure-oriented outcomes - Surgical complications in Clavien-Dindo classification | From perioperative period to post-operative 1 year
  Clavien-Dindo classification is a commonly used surgical complication grading system, from grade I-V with grade V indicating worst outcome (death).
Procedure-oriented outcomes - Completeness of lesion removal | From perioperative period to post-operative 1 year
  Indicates if the vocal fold pathology has been completely removed
Procedure-oriented outcomes - Operation time | From perioperative period to post-operative 1 year
  Comparison of the operation time between two groups in terms of minute.
Patient-oriented outcomes | Perioperative period
  Patient-oriented outcomes included peri-operative throat, nose, and overall discomfort in visual analogue scale, a 10-point scale with 0 (least uncomfortable) to 10 (most uncomfortable).
Medical costs | From enrolment to post-operative 1year
  Medical costs of both interventions would be also calculated respectively, including costs for inpatient hospital stay, medical staff, operating theater and consumable.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misono S, Yueh B, Stockness AN, House ME, Marmor S. Minimal Important Difference in Voice Handicap Index-10. JAMA Otolaryngol Head Neck Surg. 2017 Nov 1;143(11):1098-1103. doi: 10.1001/jamaoto.2017.1621. PMID 28973078
- [Background] Ng E, Law T, Tang EC, Ho FN, Tong MC, Lee KY. The Cutoff Point and Diagnostic Accuracy of the Voice Handicap Index in Cantonese-Speaking Population. J Voice. 2021 Mar;35(2):163-168. doi: 10.1016/j.jvoice.2020.09.021. Epub 2020 Oct 9. PMID 33046276
- [Background] Gao WZ, Abu-Ghanem S, Reder LS, Amin M, Johns MM. A Novel Approach to Vocal Fold Mucous Retention Cysts: Awake KTP Laser-Assisted Marsupialization. J Voice. 2022 Jul;36(4):570-573. doi: 10.1016/j.jvoice.2020.07.028. Epub 2020 Aug 22. PMID 32843259
- [Background] Gocal WA, Tong JY, Maxwell PJ, Sataloff RT. Systematic Review of Recurrence Rates of Benign Vocal Fold Lesions Following Surgery. J Voice. 2025 May;39(3):787-798. doi: 10.1016/j.jvoice.2022.10.015. Epub 2022 Dec 10. PMID 36513559
- [Background] Hsu CM, Armas GL, Su CY. Marsupialization of vocal fold retention cysts: voice assessment and surgical outcomes. Ann Otol Rhinol Laryngol. 2009 Apr;118(4):270-5. doi: 10.1177/000348940911800406. PMID 19462847
- [Background] Courey MS, Gardner GM, Stone RE, Ossoff RH. Endoscopic vocal fold microflap: a three-year experience. Ann Otol Rhinol Laryngol. 1995 Apr;104(4 Pt 1):267-73. doi: 10.1177/000348949510400402. PMID 7717615
- [Background] Tam AKY, Leung NMW, Lee SKJ, Wei Y, Hu Y, Chan JYK, Law T. Randomized Controlled Trial of Awake Transnasal Laser-Assisted Surgery for Benign Laryngeal Lesions. Laryngoscope. 2024 Aug;134(8):3732-3740. doi: 10.1002/lary.31481. Epub 2024 May 10. PMID 38727019
- [Background] Schimberg AS, Wellenstein DJ, van den Broek EM, Honings J, van den Hoogen FJA, Marres HAM, Takes RP, van den Broek GB. Office-based vs. operating room-performed laryngopharyngeal surgery: a review of cost differences. Eur Arch Otorhinolaryngol. 2019 Nov;276(11):2963-2973. doi: 10.1007/s00405-019-05617-z. Epub 2019 Sep 5. PMID 31486936
- [Background] Lin YH, Wang CT, Lin FC, Liao LJ, Lo WC, Cheng PW. Treatment Outcomes and Adverse Events Following In-Office Angiolytic Laser With or Without Concurrent Polypectomy for Vocal Fold Polyps. JAMA Otolaryngol Head Neck Surg. 2018 Mar 1;144(3):222-230. doi: 10.1001/jamaoto.2017.2899. PMID 29346486
- [Background] Wellenstein DJ, Honings J, Schimberg AS, Schutte HW, Herruer JM, van den Hoogen FJA, Takes RP, van den Broek GB. Office-based CO2 laser surgery for benign and premalignant laryngeal lesions. Laryngoscope. 2020 Jun;130(6):1503-1507. doi: 10.1002/lary.28278. Epub 2019 Sep 9. PMID 31498454
- [Background] Shoffel-Havakuk H, Sadoughi B, Sulica L, Johns MM 3rd. In-office procedures for the treatment of benign vocal fold lesions in the awake patient: A contemporary review. Laryngoscope. 2019 Sep;129(9):2131-2138. doi: 10.1002/lary.27731. Epub 2018 Dec 21. PMID 30575043

DOCUMENTS (1):
  • Study Protocol (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT06703515/Prot_000.pdf